CLINICAL TRIAL: NCT00219804
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Tetrabenazine for the Treatment of Huntington's Chorea
Brief Title: Efficacy and Safety of Tetrabenazine in Chorea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prestwick Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 103,004
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2005-09

CONDITIONS: Huntington's Disease
MeSH Terms: conditions — Huntington Disease | interventions — Tetrabenazine

INTERVENTIONS:
Drug: tetrabenazine or placebo

SUMMARY:
The primary objective of this study was to establish the absolute reduction of chorea in participants with Huntington's disease(HD) treated with tetrabenazine or placebo

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* suffer from manifest HD as confirmed by genetic testing
* Meet chorea and total functional capacity scores on Unified Huntington's Disease Rating Scale
* Meet criteria on Hamilton Depression Rating Scale, Unified Parkinson's Disease Rating Scale dysphagia and dysarthria scale
* Independently ambulatory

Exclusion Criteria

* previous treatment with tetrabenazine
* unstable or serious medical or psychiatric illness
* concomitant use identified drugs
* untreated depression
* lack of caregiver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Fred Marshall, M.D., Principal Investigator — Huntington's Study Group

REFERENCES:
- [Derived] Claassen DO, Carroll B, De Boer LM, Wu E, Ayyagari R, Gandhi S, Stamler D. Indirect tolerability comparison of Deutetrabenazine and Tetrabenazine for Huntington disease. J Clin Mov Disord. 2017 Mar 1;4:3. doi: 10.1186/s40734-017-0051-5. eCollection 2017. PMID 28265459
- [Derived] Frank S. Tetrabenazine as anti-chorea therapy in Huntington disease: an open-label continuation study. Huntington Study Group/TETRA-HD Investigators. BMC Neurol. 2009 Dec 18;9:62. doi: 10.1186/1471-2377-9-62. PMID 20021666